CLINICAL TRIAL: NCT04843462
Title: A Randomized, Controlled Pragmatic Trial Assessing the Value of an add-on Therapy With Edupression.Com® in Therapy Resistant Depressive Patients Treated With Esketamine Nasal Spray
Brief Title: Add-on Therapy With Edupression.Com® on Therapy Resistant Depressive Patients Treated With Nasal Esketamine Spray
Acronym: Esketamin+
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lukas Pezawas (Other)
Responsible Party: Sponsor-Investigator, Lukas Pezawas, Assoc.Prof. Priv.Doz. Dr. Lukas Pezawas, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2467/2020
Record Dates: First submitted 2021-04-07; First posted 2021-04-13 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Major Depressive Disorder; Therapy Resistant Depression
Keywords: Depression; Esketamine; Treatment resistant depression; Internet-based intervention; Telemedicine
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant; Depression

STUDY DESIGN:
Intervention Model Description: The interventional study consists of two parallel study arms. The interventional group receives "treatment-as-usual" with nasal esketamine spray and access to edupression.com®. The control group only receives "treatment-as-usual".
Who Masked: Participant
Masking Description: Data will be immediately pseudonymized and stored as a master list at the internal server of the MUV (Medical University Vienna). The study staff will only have access to the master list and only the principal investigator and study director will have access to the pseudonymization list. This locked place will be located at the clinic (MUV). All non-personal pseudonymized research relevant data are stored in a master list on a server of the research group at the MUV, to which study staff has access.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- edupression.com® + treatment-as-usual (Experimental): Patients are receiving treatment with edupression.com® in addition to TAU (treatment-as-usual) with esketamine nasal spray
  Interventions: Device: edupression.com®; Drug: Esketamine nasal spray
- treatment-as-usual (Active Comparator): Patients are receiving TAU (treatment-as-usual) with esketamine nasal spray
  Interventions: Drug: Esketamine nasal spray

INTERVENTIONS:
Device: edupression.com® — Edupression.com® is an evidence-based self-help program that was developed for the treatment of mild to moderate unipolar depression. It is based on two core foundations, psychoeducation with elements of cognitive behavior therapy (CBT) and a mood chart. Both foundations are registered as a medical product. As such, detailed risk management documentation includes probability and severity of adverse events. Moreover, detailed strategies such as warnings were implemented in the software and documented accordingly.
  It can be used on a PC as well as on mobile devices (browser, app) at any time.
  Arms: edupression.com® + treatment-as-usual
Drug: Esketamine nasal spray — All patients included in this study are receiving esketamine nasal spray as treatment-as-usual

SUMMARY:
Pragmatic clinical trial of an add-on therapy regarding the use of edupression.com® - a licensed computer based self-help program - on patients with therapy-resistant depression receiving esketamine nasal spray

DETAILED DESCRIPTION:
edupression.com® - is a medical product and computer based self-help program based on cognitive behavioral therapy, psychoeducation and mood tracking. Patients included in the interventional arm of this study are receiving full access to edupression.com®.

Due to limited resources regarding face-to-face therapy and a high prevalence of Major Depressive Disorder - of which 37% can be identified as therapy-resistant depression (TRD) according to the definition of the European Medical Agency (EMA) - low-intensity psychosocial interventions such as edupression.com® are recommended as first-line digital therapeutic agent by international guidelines such as National Institute for Health and Care Excellence (NICE) guidelines. Studies have shown that digital interventions - such as edupression.com - show comparable clinical efficiency to face-to-face therapy and therefore could be able to fill the gap in limited ressources. In this study patients with therapy-resistant depression are receiving therapy with edupression.com® in addition to their treatment-as-usual with esketamine nasal spray. Comparable studies have shown that patients receiving psychotherapy in addition to their medical therapy benefit in regards to their clinical outcome. Considering these findings, this study is aimed to investigate potential clinical benefits in patients receiving digital therapy with edupression®.com as an add-on therapy to their treatment-as-usual therapy with esketamine nasal spray.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Initial MADRS-Score of 22 or above
* Diagnosis of a therapy-resistant depression following the definition of the European Medicines Agency (EMA) - absence of remission after two or more guideline-oriented therapies
* Patients assigned to treatment with nasal esketamine spray Spravato®
* Signed informed consent
* Native German speaker
* Basic knowledge in using computers/smartphones operationalized as daily use of at least two devices (such as tablets, computers, smartphones etc)

Exclusion Criteria:

* Contraindication regarding the use of Spravato®
* Diagnosis of one of the following psychiatric comorbidities: substance abuse, schizoaffective disorders, schizophrenia, bipolar disorder, organic disorders diagnosed via Mini International Neuropsychiatric Interview (MINI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-04-29 (Actual); Primary Completion 2023-04-14 (Estimated); Study Completion 2023-04-14 (Estimated)

PRIMARY OUTCOMES:
Therapy response (observer-rated) | At week 4, 8 and 12 after baseline
  Change in depressive symptoms according to MADRS-Score (0-60 points, higher values stand for)
Percentage of received esketamine treatments in relation to scheduled ones | Percentage of received esketamine treatments in relation to scheduled ones after 12 weeks
  Change in therapy adherence according to a percentual increase of received esketamine treatments in accordance to scheduled ones

SECONDARY OUTCOMES:
Therapy response (self-rated) | At week 4, 8 and 12 after baseline
  Change in depressive symptoms according to the self rating scale PHQ-9 (Patient Health Questionnaire-9) (1-27 points, higher values stand for increased severity)

CONTACTS AND LOCATIONS:
Overall Officials: Markus Dold, MD., Priv.Doz., Study Chair — Medical University of Vienna; Gabriele Fischer, MD, Prof., Study Chair — Medical University of Vienna; Lukas M Pezawas, MD, Prof., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] National Collaborating Centre for Mental Health (UK). Depression: The Treatment and Management of Depression in Adults (Updated Edition). Leicester (UK): British Psychological Society; 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK63748/ PMID 22132433
- [Result] Luo C, Sanger N, Singhal N, Pattrick K, Shams I, Shahid H, Hoang P, Schmidt J, Lee J, Haber S, Puckering M, Buchanan N, Lee P, Ng K, Sun S, Kheyson S, Chung DC, Sanger S, Thabane L, Samaan Z. A comparison of electronically-delivered and face to face cognitive behavioural therapies in depressive disorders: A systematic review and meta-analysis. EClinicalMedicine. 2020 Jun 27;24:100442. doi: 10.1016/j.eclinm.2020.100442. eCollection 2020 Jul. PMID 32775969